CLINICAL TRIAL: NCT04272736
Title: Evaluating the Compliance, Acceptability, Safety and Tolerance of a Lower Calorie Protein Substitute for the Dietary Management of Phenylketonuria in Children and Adults - a Pilot Study
Brief Title: PKU Low Calorie Drink Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not started, not funded
Sponsor: Nutricia UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PKULite2018
Record Dates: First submitted 2018-08-29; First posted 2020-02-17 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Phenylketonurias; Hyperphenylalaninaemia
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Low calorie protein substitute (Experimental): Single arm designed, 3 day baseline, 28 day on the lower calorie amino acid based liquid protein substitute.
  Interventions: Dietary Supplement: Low calorie protein substitute

INTERVENTIONS:
Dietary Supplement: Low calorie protein substitute — The evaluated dietary supplement is a lower calorie amino acid based liquid protein substitute designed for patients with PKU.

SUMMARY:
This study will evaluate the compliance, acceptability, gastrointestinal (GI) tolerance and safety of a lower calorie amino acid based liquid protein substitute for patients with Phenylketonuria (PKU) or hyperphenylalaninemia (HPA).

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 3 years of age or above
* Diagnosed with classical or variant type phenylketonuria (PKU), or hyperphenylalaninemia (HPA)
* Have been compliant in taking at least one amino acid-based, Phe-free protein substitute, providing at least 20g protein equivalent daily, for at least 1 month prior to study commencement
* Have a prescribed daily Phe allowance
* Written informed consent from patient, or from parent / carer if applicable

Exclusion Criteria:

* Pregnant or lactating
* Requiring enteral tube or parenteral nutrition
* Major hepatic or renal dysfunction
* Participation in other studies within 1 month prior to entry to this study
* Allergy to any of the study product ingredients
* Investigator concern around the patient being underweight (e.g.: BMI lower than 18.5kg/m2 for adults) and/or having an eating disorder
* Investigator concern around willingness/ability of patient or parent/carer to comply with protocol requirements

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Compliance | Daily for 31 days
  Questionnaire on amounts offered and amounts actually consumed, compared to recommended amount. Amounts (values) are recorded

SECONDARY OUTCOMES:
Acceptability: Tick-box questionnaire | Recorded at baseline and end of intervetnion (day 31)
  Tick-box questionnaire on overall liking and acceptability of product (ie dislike a lot, dislike moderately, neutral, like moderately, like a lot)
Blood phenylalanine and other amino acid levels | Recorded at baselien and end of intervention (day 31)
  Blood spot test.
Gastro-intestinal tolerance | recorded at baseline, beginning of intervention and end of intervention(12 out of 31 days in total)
  Questionnaire detailing any GI symptoms, severity (none, mild, moderate, severe) and change from usual.
Nutrient intake | Recorded at basleine and end of intervention (day 31)
  24h dietary recall.
Anthropometry | Recorded at baseline and end of intervention (day 31)
  Measurements of height (m) and weight (kg) at baseline and end of study.

IPD SHARING:
Plan to Share IPD: No